CLINICAL TRIAL: NCT04975412
Title: Relationship of Whole Blood Zinc Levels to Acne Severity Among Filipinos 18-25 Years Old: A Cross-sectional Comparative Study
Brief Title: Relationship of Whole Blood Zinc Levels to Acne Severity
Status: Completed | Type: Observational
Sponsor: East Avenue Medical Center, Philippines (Other Government)
Responsible Party: Principal Investigator, Monique Lianne C. Lim-Ang, MD, MBA, DPDS, Principal Investigator, East Avenue Medical Center, Philippines
Other Study IDs: EAMC IERB 2017-40
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Zinc in blood; Global Acne Grading System
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acne vulgaris group (cases): Filipino patients, aged 18-25 years old with diagnosis of Acne Vulgaris
  Interventions: Diagnostic Test: Whole blood zinc level
- control group: healthy Filipino patients, aged 18-25 years old
  Interventions: Diagnostic Test: Whole blood zinc level

INTERVENTIONS:
Diagnostic Test: Whole blood zinc level — whole blood zinc levels determined through ashing acid digestion-inductively coupled plasma (ICP) using Shimadzu ICPS-7510, an inductively coupled plasma emission spectrometer.

SUMMARY:
Acne Vulgaris is one of the most common dermatologic diagnoses in the world. A number of studies have been conducted comparing serum zinc levels with acne vulgaris; however, no studies have yet been done in the Philippine setting.

The objective of this study is to determine the relationship between whole blood zinc levels and the severity of acne vulgaris in Filipino patients and normal controls who are 18-25 years old.

DETAILED DESCRIPTION:
Acne Vulgaris is a disorder of the pilosebaceous unit characterized by formation of comedones, papules, pustules, inflamed nodules, and cysts.1 Most common predilection sites are those with hormonally sensitive sebaceous glands such as the face, neck, chest, upper back and upper arms. Acne can persist for years and result in disfigurement and permanent scarring. It can cause serious adverse effects on psychosocial development, resulting in emotional problems, withdrawal from society, and depression. Nearly all adolescents experience different severity levels of acne vulgaris, with moderate to severe levels affecting around 20% of this population. In the Philippines, high school students were found to have a mild impairment of quality of life (QOL) due to acne, regardless of severity. Despite the known treatment regimens for acne, people are still suffering from the effects of the disease.

Acne has four main pathogenic contributors: follicular hyperkeratinization, increased sebum production, Propionibacterium acnes (P. acnes) within the follicle, and inflammation. Reports show that antibiotic resistance is a growing issue in the treatment regimen of acne vulgaris, making it less and less suitable for long-term treatment. Other options that can be substitutes or adjuncts to treatment may be useful in this condition.

Zinc is an essential element for normal epithelial differentiation and for normal development. It has also been shown to have antioxidant properties. At present, there is paucity of data regarding the role of zinc levels in the development or severity of acne vulgaris. Also, data on favorable effects of dietary factors such as zinc, omega-3 fatty acids, antioxidants, vitamin A, and dietary fiber on acne vulgaris are limited specially in the Philippines.

This study will be conducted to measure the whole blood zinc levels in patients with acne vulgaris and compare it with healthy controls. This aims to determine the relationship between whole blood zinc levels and disease severity in Filipino patients with acne vulgaris in order to bring new insight to guide further studies regarding zinc's role in the pathogenesis and possible further treatment of acne vulgaris in the Philippines.

Significance of the Study:

While a number of studies have been conducted comparing serum zinc levels with acne vulgaris, no previous studies have been done in the Philippine setting that assesses the relationship of whole blood zinc levels with the severity of acne. Given that acne vulgaris is one of the most common dermatologic diagnoses in the Philippine population, and the increasing resistance to antibiotics commonly used to treat acne, studies about other treatment modalities for acne vulgaris that do not have resistance factors are timely and significant in the country.

For long-term or maintenance therapy, physicians should consider effectivity, cost, and adverse effects. By determining the relationship of whole blood zinc levels to acne severity among Filipinos 18-25 years old, this study can be used as evidence for giving zinc supplements to Filipino people diagnosed with acne vulgaris if a significant relationship is found. Since zinc is more cost-effective and has less adverse effects compared to most antibiotics, this may prove helpful for the Filipino patient in terms of safety and economy for long-term therapy. Furthermore, this study may also be able to provide more information for further studies towards non-antimicrobial treatment regimens for acne vulgaris in the Philippines.

Research Question:

Is there a relationship between whole blood zinc levels and the severity of acne vulgaris in Filipino patients 18-25 years old versus normal controls?

Null Hypothesis: There is no relationship between whole blood zinc levels and the severity of acne vulgaris.

Alternative Hypothesis: There is a relationship between whole blood zinc levels and the severity of acne vulgaris.

Objectives:

* To study the relationship between whole blood zinc levels and the severity of acne vulgaris in Filipino patients 18-25 years old and normal controls
* To describe the clinical profile of Filipino patients 18-25 years old with acne vulgaris
* To determine the whole blood zinc levels of acne patients compared to controls
* To determine the relationship of the clinical severity of acne vulgaris to whole blood zinc levels

A cross-sectional comparative study design will be utilized for this study which will be conducted from November 2017 to March 2018. The study will be conducted at the Dermatology Out-patient Clinic of the East Avenue Medical Center (EAMC).

STUDY PROCEDURE

1. The study will be submitted to the Technical Review Board and Institution Ethics and Review Board for approval.
2. In the Dermatology Out-Patient Department of East Avenue Medical Center, patients seeking consult for their skin lesions which were diagnosed to be Acne Vulgaris will be screened if they meet the inclusion/exclusion criteria.
3. Informed consent will be obtained for those who are qualified.
4. Patients will be given proper treatment whether they agree to participate or not. For the patients who agree to participate, the investigator will assess the patient's acne severity using the Global Acne Grading Scale (GAGS).
5. Twelve milliliters of blood will be extracted from the patient with proper aseptic technique and waste disposal.
6. Blood sample will be properly stored in three EDTA tubes, labelled, and transported to the laboratory for determination of whole blood zinc levels through ashing acid digestion- inductively coupled plasma (ICP) using Shimadzu ICPS-7510, an inductively coupled plasma emission spectrometer.

   1. Blood samples are viable and stable for 5 days at 15-25 degrees Celsius.
   2. A memorandum of agreement between the principal investigator and Hi-Precision Diagnostics, Inc. has been made. Hi-Precision Diagnostics will be providing the materials for extraction, picking-up, and transporting the blood sample using a special insulated medical specimen bag (Versapak Pathology and Specimen bag) with ice packs and thermometer to help maintain the ideal temperature of 15-25 degrees Celsius.
   3. Schedule of specimen pick-up is from 8:00 am- 8:00 pm and may be done on an as-needed basis. The blood specimens will be stored in the refrigerator immediately after extraction.
7. Results will be obtained by the investigator via the online results portal of the laboratory.
8. Data collected will be tabulated and data analysis will be done.

PASS 2008 was used for the computation of minimum sample size. Parameters for the computation was obtained from previously published studies. For the one-way ANOVA, a minimum of 40 patients (10 for each acne severity: mild, moderate and severe acne and 10 for controls) achieves 95% power to detect differences among the means versus the alternative of equal means using an F test with a significance level of 0.05. The size of the variation in the means is represented by their standard deviation which is 13.30 mg/dL and the common standard deviation within a group is assumed to be 20.00 mg/dL.

Data will be encoded by the researcher in MS Excel. The excel file will be converted into Stata file for further data processing and analysis. Stata SE version 12 will be used for both descriptive and inferential statistics. Quantitative variables will be presented as mean or median while qualitative variables will be presented as percentages.

In order to compare the whole blood zinc levels between cases and controls, independent T-test will be used. ANOVA will be used to compare the whole blood zinc levels by acne severity. Multiple linear regression analysis will then be performed in order to determine the association of whole blood zinc levels with acne severity after controlling for the effects of significant confounding variables. All p values ≤ 0.05 will be considered as significant.

The correlation of whole blood zinc levels with severity of acne vulgaris in Filipino patients may help clinicians recommend more detailed dietary advice and add non-antibiotic supplements to their current treatment of acne vulgaris. The results of the study can serve as a guide for further studies related to whole blood zinc and its role in the pathogenesis of acne vulgaris in Filipino patients.

ELIGIBILITY:
Inclusion Criteria for cases:

* Filipino patients, aged 18-25 years old
* Diagnosis of acne vulgaris
* Able to read and write in English or Tagalog
* Seen at the dermatology out-patient department of East Avenue Medical Center

Exclusion Criteria for cases:

* Patients with other chronic dermatoses or systemic disease
* Taking oral supplements or medications for the past 3 months
* Patients who are pregnant or lactating

Inclusion Criteria for controls:

* Filipino patients, aged 18-25 years old
* Able to read and write in English or Tagalog
* Seen at the dermatology out-patient department of East Avenue Medical Center

Exclusion Criteria for controls:

* Patients with acne vulgaris or other chronic dermatoses or systemic disease
* Taking oral supplements or medications for the past 3 months
* Patients who are pregnant or lactating

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects of the study included patients clinically diagnosed with acne vulgaris and healthy controls, aged 18-25 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Acne severity | initial consult
  Based on the Global Acne Grading System (GAGS) score. Minimum value 0, maximum value 44. Acne severity is rated as mild (1-18), moderate (19-30), severe (31-38), and very severe (≥39). Control patients have GAGS score of 0.
Whole blood zinc level | initial consult
  whole blood zinc level in µg/mL

SECONDARY OUTCOMES:
demographics | initial consult
  age and sex

CONTACTS AND LOCATIONS:
Overall Officials: Monique Lianne C. Lim-Ang, MD,MBA,DPDS, Principal Investigator — East Avenue Medical Center
Locations (1):
- East Avenue Medical Center, Quezon City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhate K, Williams HC. Epidemiology of acne vulgaris. Br J Dermatol. 2013 Mar;168(3):474-85. doi: 10.1111/bjd.12149. PMID 23210645
- [Background] Prasad AS. Zinc is an Antioxidant and Anti-Inflammatory Agent: Its Role in Human Health. Front Nutr. 2014 Sep 1;1:14. doi: 10.3389/fnut.2014.00014. eCollection 2014. PMID 25988117
- [Background] Tan JK, Bhate K. A global perspective on the epidemiology of acne. Br J Dermatol. 2015 Jul;172 Suppl 1:3-12. doi: 10.1111/bjd.13462. PMID 25597339
- [Background] Collier CN, Harper JC, Cafardi JA, Cantrell WC, Wang W, Foster KW, Elewski BE. The prevalence of acne in adults 20 years and older. J Am Acad Dermatol. 2008 Jan;58(1):56-9. doi: 10.1016/j.jaad.2007.06.045. Epub 2007 Oct 22. PMID 17945383
- [Background] Goulden V, Stables GI, Cunliffe WJ. Prevalence of facial acne in adults. J Am Acad Dermatol. 1999 Oct;41(4):577-80. PMID 10495379
- [Background] Humphrey S. Antibiotic resistance in acne treatment. Skin Therapy Lett. 2012 Oct;17(9):1-3. PMID 23032935
- [Background] Al-Shobaili HA. Oxidants and anti-oxidants status in acne vulgaris patients with varying severity. Ann Clin Lab Sci. 2014 Spring;44(2):202-7. PMID 24795060
- [Background] Rostan EF, DeBuys HV, Madey DL, Pinnell SR. Evidence supporting zinc as an important antioxidant for skin. Int J Dermatol. 2002 Sep;41(9):606-11. doi: 10.1046/j.1365-4362.2002.01567.x. PMID 12358835
- [Background] Buxaderas SC, Farre-Rovira R. Whole blood and serum zinc levels in relation to sex and age. Rev Esp Fisiol. 1985 Dec;41(4):463-70. PMID 4095368
- [Background] Rostami Mogaddam M, Safavi Ardabili N, Maleki N, Soflaee M. Correlation between the severity and type of acne lesions with serum zinc levels in patients with acne vulgaris. Biomed Res Int. 2014;2014:474108. doi: 10.1155/2014/474108. Epub 2014 Jul 24. PMID 25157359
- [Background] Michaelsson G, Vahlquist A, Juhlin L. Serum zinc and retinol-binding protein in acne. Br J Dermatol. 1977 Mar;96(3):283-6. doi: 10.1111/j.1365-2133.1977.tb06138.x. PMID 139912
- [Background] Adityan B, Kumari R, Thappa DM. Scoring systems in acne vulgaris. Indian J Dermatol Venereol Leprol. 2009 May-Jun;75(3):323-6. doi: 10.4103/0378-6323.51258. No abstract available. PMID 19439902
- [Background] Ozuguz P, Dogruk Kacar S, Ekiz O, Takci Z, Balta I, Kalkan G. Evaluation of serum vitamins A and E and zinc levels according to the severity of acne vulgaris. Cutan Ocul Toxicol. 2014 Jun;33(2):99-102. doi: 10.3109/15569527.2013.808656. Epub 2013 Jul 5. PMID 23826827
- [Background] Ikaraoha CI, Mbadiwe NC, Anyanwu CJ, Odekhian J, Nwadike CN, Amah HC. The Role of Blood Lead, Cadmium, Zinc and Copper in Development and Severity of Acne Vulgaris in a Nigerian Population. Biol Trace Elem Res. 2017 Apr;176(2):251-257. doi: 10.1007/s12011-016-0839-4. Epub 2016 Sep 6. PMID 27600928
- [Background] Amer M, Bahgat MR, Tosson Z, Abdel Mowla MY, Amer K. Serum zinc in acne vulgaris. Int J Dermatol. 1982 Oct;21(8):481-4. doi: 10.1111/j.1365-4362.1982.tb03188.x. PMID 6217164
- [Background] Arora PN, Dhillon KS, Rajan SR, Sayal SK, Das AL. Serum Zinc Levels in Cutaneous Disorders. Med J Armed Forces India. 2002 Oct;58(4):304-6. doi: 10.1016/S0377-1237(02)80083-1. Epub 2011 Jul 21. PMID 27407419
- [Background] Canavan TN, Chen E, Elewski BE. Optimizing Non-Antibiotic Treatments for Patients with Acne: A Review. Dermatol Ther (Heidelb). 2016 Dec;6(4):555-578. doi: 10.1007/s13555-016-0138-1. Epub 2016 Aug 19. PMID 27541148
- [Background] Gupta M, Mahajan VK, Mehta KS, Chauhan PS. Zinc therapy in dermatology: a review. Dermatol Res Pract. 2014;2014:709152. doi: 10.1155/2014/709152. Epub 2014 Jul 10. PMID 25120566
- [Background] Sardana K, Chugh S, Garg VK. The role of zinc in acne and prevention of resistance: have we missed the "base" effect? Int J Dermatol. 2014 Jan;53(1):125-7. doi: 10.1111/ijd.12264. No abstract available. PMID 24350859
- [Background] Bray TM, Bettger WJ. The physiological role of zinc as an antioxidant. Free Radic Biol Med. 1990;8(3):281-91. doi: 10.1016/0891-5849(90)90076-u. PMID 2187766
- [Background] Lim KH, Riddell LJ, Nowson CA, Booth AO, Szymlek-Gay EA. Iron and zinc nutrition in the economically-developed world: a review. Nutrients. 2013 Aug 13;5(8):3184-211. doi: 10.3390/nu5083184. PMID 23945676
- [Background] Plum LM, Rink L, Haase H. The essential toxin: impact of zinc on human health. Int J Environ Res Public Health. 2010 Apr;7(4):1342-65. doi: 10.3390/ijerph7041342. Epub 2010 Mar 26. PMID 20617034
- [Background] Oteiza PI. Zinc and the modulation of redox homeostasis. Free Radic Biol Med. 2012 Nov 1;53(9):1748-59. doi: 10.1016/j.freeradbiomed.2012.08.568. Epub 2012 Aug 25. PMID 22960578
- [Background] Maret W. Zinc biochemistry: from a single zinc enzyme to a key element of life. Adv Nutr. 2013 Jan 1;4(1):82-91. doi: 10.3945/an.112.003038. PMID 23319127
- [Background] Rangan AM, Samman S. Zinc intake and its dietary sources: results of the 2007 Australian National Children's Nutrition and Physical Activity Survey. Nutrients. 2012 Jul;4(7):611-24. doi: 10.3390/nu4070611. Epub 2012 Jun 26. PMID 22852053
- [Background] Toyoda M, Morohashi M. Pathogenesis of acne. Med Electron Microsc. 2001 Mar;34(1):29-40. doi: 10.1007/s007950100002. PMID 11479771
- [Background] Aydemir EH. Acne vulgaris. Turk Pediatri Ars. 2014 Mar 1;49(1):13-6. doi: 10.5152/tpa.2014.1943. eCollection 2014 Mar. PMID 26078626
- [Background] Akhtar S. Zinc status in South Asian populations--an update. J Health Popul Nutr. 2013 Jun;31(2):139-49. doi: 10.3329/jhpn.v31i2.16378. PMID 23930332
- [Background] Eady EA, Gloor M, Leyden JJ. Propionibacterium acnes resistance: a worldwide problem. Dermatology. 2003;206(1):54-6. doi: 10.1159/000067822. PMID 12566805
- [Background] Eady EA, Cove JH, Holland KT, Cunliffe WJ. Erythromycin resistant propionibacteria in antibiotic treated acne patients: association with therapeutic failure. Br J Dermatol. 1989 Jul;121(1):51-7. doi: 10.1111/j.1365-2133.1989.tb01399.x. PMID 2527056
- [Background] Ross JI, Snelling AM, Carnegie E, Coates P, Cunliffe WJ, Bettoli V, Tosti G, Katsambas A, Galvan Perez Del Pulgar JI, Rollman O, Torok L, Eady EA, Cove JH. Antibiotic-resistant acne: lessons from Europe. Br J Dermatol. 2003 Mar;148(3):467-78. doi: 10.1046/j.1365-2133.2003.05067.x. PMID 12653738
- [Background] Cooper AJ. Systematic review of Propionibacterium acnes resistance to systemic antibiotics. Med J Aust. 1998 Sep 7;169(5):259-61. doi: 10.5694/j.1326-5377.1998.tb140250.x. PMID 9762064
- [Background] Leyden JJ, McGinley KJ, Cavalieri S, Webster GF, Mills OH, Kligman AM. Propionibacterium acnes resistance to antibiotics in acne patients. J Am Acad Dermatol. 1983 Jan;8(1):41-5. doi: 10.1016/s0190-9622(83)70005-8. PMID 6219134
- See also: Toxicological profile for zinc — http://www.atsdr.cdc.gov/toxprofiles/tp60-c7.pdf
- See also: Serum Trace Elements (Zinc, Copper and Magnesium) Status in Iraqi Patients with Acne Vulgaris:( Case- Controlled Study) — http://www.iasj.net/iasj/download/0354b90b97bd276f
- See also: Zinc Levels in Patients with Acne Vulgaris — http://jtad.org/archives/archive-detail/article-preview/zinc-levels-in-patients-with-acne-vulgaris/32246
- See also: Effect of Serum Trace Elements, Macro-minerals and Antioxidants in Acne Vulgaris Patients: A Case-Control Study — http://www.banglajol.info/index.php/JPharma/article/view/30940

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT04975412/Prot_SAP_000.pdf